CLINICAL TRIAL: NCT03400384
Title: Using Policy to Reduce Opioids by Educating and Empowering Patients With Chronic Non-cancer Pain: The TAPERING Randomised Trial.
Brief Title: Trial Applying Policy to Eliminate or Reduce Inappropriate Narcotics in the General-population
Acronym: TAPERING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Cara Tannenbaum, Professor in the faculties of Medicine and Pharmacy, University of Montreal, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CIHR 201506PHSI-337814-MB
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Inappropriate Dose of Drug Administered; Pain, Chronic; Health Behavior
Keywords: Deprescribing
MeSH Terms: conditions — Chronic Pain; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct-to-consumer educational brochure (Experimental): The intervention arm will be mailed an evidence-based, theory-driven direct-to-consumer educational brochure, highlighting the potential benefits and harms of opioids when used to treat chronic non-cancer pain.
  Interventions: Other: Direct-to-consumer educational brochure
- Control wait list (No Intervention): This arm will receive the intervention at the completion of the six-month follow-up period for the intervention group.

INTERVENTIONS:
Other: Direct-to-consumer educational brochure — The intervention arm will be mailed an evidence-based, theory-driven direct-to-consumer educational brochure, highlighting the potential benefits and harms of opioids when used to treat chronic non-cancer pain.
  Arms: Direct-to-consumer educational brochure

SUMMARY:
To assess the effectiveness of a government-led population-based opioid intervention on discontinuation of opioid medication in community-dwelling adults with chronic non-cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults registered to receive pharmaceutical benefits in Manitoba, who are aged 18 years and over and who have received ≥90 days supply of opioids in the 6 months prior to the trial will be included. This will ensure chronic use and episodic use of opioids will be included.

Exclusion Criteria:

* People receiving palliative care, people with cancer, and people who receive opioids in hospital. People with dementia (identified by having received a prescription for memantine or a cholinersterase inhibitor in the previous 12 months) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4255 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Complete cessation of opioids | 6 months
  Provincial prescription insurance claims will be used to measure whether or not opioids are dispensed to community-dwelling adults randomized to either the intervention or control groups between baseline and 6-month follow up. Prescription data contain information on all dispensed prescriptions including drug name, dispensing date, dosage, drug form, the quantity of the drug dispensed, and the license number of the physician who wrote the prescription. Discontinuation of an opioid will be defined as the lack of a prescription claim for at least 60 days.

SECONDARY OUTCOMES:
Dose reduction or therapeutic switch to an alternate analgesic | 6 months
  The magnitude and direction of dose changes will be assessed for people who do not achieve the primary endpoint of complete cessation. New pharmacy dispensing of a prescription for a lower strength, or supply of a reduced quantity of tablets/patches will be considered in the dose reduction calculation. Where substitution to an alternative opioid occurs, opioid doses will be converted to "oral morphine equivalents" to determine the magnitude and direction of the change. A therapeutic switch will be indicated by a new dispensing for an alternative medication class.
The proportion of people achieving opioid doses below 90mg oral morphine equivalents. | 6 months
  All opioids will be converted to an oral morphine equivalent dose. The proportion of patients who are prescribed <90mg of oral morphine equivalent at the end of the 6-month follow up will be compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Tannenbaum, MD, MSc, Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (1):
- Institut universitaire de gériatrie de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner JP, Halme AS, Caetano P, Langford A, Tannenbaum C. Government Direct-to-Consumer Education to Reduce Prescription Opioid Use: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2413698. doi: 10.1001/jamanetworkopen.2024.13698. PMID 38809554
- [Derived] Turner JP, Caetano P, Tannenbaum C. Leveraging policy to reduce chronic opioid use by educating and empowering community dwelling adults: a study protocol for the TAPERING randomized controlled trial. Trials. 2019 Jul 9;20(1):412. doi: 10.1186/s13063-019-3508-z. PMID 31288859